CLINICAL TRIAL: NCT00000191
Title: Carbamazepine Treatment for Cocaine Dependence
Brief Title: Carbamazepine Treatment for Cocaine Dependence - 5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, James Cornish, Principal Investigator, University of Pennsylvania
Purpose: Treatment
Other Study IDs: NIDA-00144-5; 3R01DA012268 (NIH); K20-00144-5
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Cocaine-Related Disorders
Keywords: Cocaine Dependence; Carbamazepine
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Carbamazepine

INTERVENTIONS:
Drug: Carbamazepine

SUMMARY:
The purpose of this study is to assess carbamazepine as a pharmacotherapy for cocaine dependence.

ELIGIBILITY:
Please contact site for information.

Ages: 21 Years to 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1991-01; Primary Completion 1994-02 (Actual); Study Completion 1994-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Cornish, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Cornish JW, Maany I, Fudala PJ, Neal S, Poole SA, Volpicelli P, O'Brien CP. Carbamazepine treatment for cocaine dependence. Drug Alcohol Depend. 1995 Jun;38(3):221-7. doi: 10.1016/0376-8716(95)01102-5. PMID 7555622